CLINICAL TRIAL: NCT05775510
Title: Study to Evaluate Neuromodulation Subject Experience With Contemporary Spinal Cord Stimulation (SCS) Modalities for Chronic Pain (SENSE SCS Clinical Study)
Brief Title: Study to Evaluate Neuromodulation Subject Experience With Contemporary Spinal Cord Stimulation (SCS) Modalities for Chronic Pain
Acronym: SENSE SCS
Status: Terminated | Type: Observational
Why Stopped: Medtronic refocused on the most impactful global evidence needs for SCS. The decision wasn't related to safety or quality. Pilot data was sufficient, but the study ended early and did not move into the Data at Scale phase.
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT22020
Record Dates: First submitted 2023-02-17; First posted 2023-03-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pain, Intractable; Pain, Chronic
MeSH Terms: conditions — Pain, Intractable; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Pilot Phase Cohort
  Interventions: Device: Commercially available neurostimulation systems
- Data at Scale Phase Cohort
  Interventions: Device: Commercially available neurostimulation systems

INTERVENTIONS:
Device: Commercially available neurostimulation systems — Spinal cord stimulation therapy delivered during trialing and following implant of commercially available neurostimulation systems

SUMMARY:
Medtronic, Inc. is sponsoring the SENSE SCS clinical study, a prospective, multi-center, post-market, non-randomized, observational study with a hybrid decentralized model of execution, utilizing a mobile application for the collection of patient reported outcomes (PROs). The purpose of the study is to evaluate workflow of a mobile application for collection of PROs and to gather data on patient experience with spinal cord stimulation therapy.

ELIGIBILITY:
Pilot Phase Inclusion Criteria:

1. 18 years of age or older
2. A clinical decision was made for the patient to receive a commercial Medtronic SCS system (trial and implant) limited to the components for an on-label indication prior to enrollment in the study. NOTE: Vectris™ SureScan™ MRI 1x8 subcompact and Specify™SureScan™ MRI 2x8 leads are not eligible system components
3. Able to differentiate between pain associated with the indication for SCS implant and other types of pain, as determined by the Investigator or designee
4. Willing and able to use a personal smart phone for study surveys. NOTE: All subjects participating in the study must be willing to download the InsightPro™ clinical trial app and maintain current software updates on their own smart phone.
5. Willing and able to provide signed and dated informed consent in English
6. Willing and able to comply with all study procedures and visits

Pilot Phase Exclusion Criteria:

1. Any active implantable neuromodulation device or system (e.g., Peripheral Nerve Stimulation, Sacral Neuromodulation)
2. Currently participating, or plans to participate, in another investigational study or has a planned major medical procedure that may interfere with study procedures or confound study results, as determined by the Investigator or designee, unless documented pre-approval is provided by the sponsor
3. Major untreated or refractory psychiatric comorbidity or other progressive disease (e.g., neurodegenerative disease, heart failure, cancer) that may confound study results, as determined by the Investigator or designee
4. Serious drug-related behavioral issues (e.g., alcohol dependency, illegal substance abuse), as determined by the Investigator or designee
5. Pregnant or planning on becoming pregnant
6. Involved in an injury claim under current litigation, beneficiary of an injury claim, or receiving worker's compensation
7. Patients with buried lead trials/implants will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended study population is adults with chronic, intractable pain of the trunk and/or limbs indicated to receive a Medtronic SCS system. Study eligibility criteria must be met to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Percentage of surveys completed from Baseline through the SCS Trial Period in the Pilot Phase Cohort. | Up to 28 days
  The percentage of surveys with complete data collected via the InsightPro™ clinical trial app from Baseline through the SCS Trial Period, calculated as the number of surveys with complete data divided by the total number of expected surveys within the Pilot Phase Cohort, expressed as a percentage.
Rating on the 7-point scale of Patient Global Impression of Change (PGIC) at Month 3 in the Data at Scale Phase Cohort | Month 3
  PGIC is a single question asking the subject to rate their improvement in pain condition on a 7-point scale from 1 (Very Much Improved) to 7 (Very Much Worse)

CONTACTS AND LOCATIONS:
Overall Officials: Mirit Argov, Study Director — Medtronic
Locations (10):
- United States (10):
  - Coastal Research Institute, Carlsbad, California
  - Pain Management Consultants of Southwest Florida, Fort Myers, Florida
  - Twin Cities Pain Clinic, Edina, Minnesota
  - Garden State Pain and Orthopedics, Clifton, New Jersey
  - Novant Health Spine Specialists, Winston-Salem, North Carolina
  - Oklahoma Pain Management, Oklahoma City, Oklahoma
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - North Texas Orthopedics and Spine Center, Grapevine, Texas
  - The San Antonio Orthopaedic Group, San Antonio, Texas
  - Procura Pain and Spine PLLC, Shenandoah, Texas